CLINICAL TRIAL: NCT05897372
Title: Feasibility of Aggressive Albuminuria Reduction in Biopsy-Proven Diabetic Nephropathy - a Pilot Study
Acronym: WP3
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Iain Bressendorff (Other)
Responsible Party: Sponsor-Investigator, Iain Bressendorff, MD PhD, Principal Investigator, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRIMETIME - WP3
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Angiotensin-Converting Enzyme Inhibitors; finerenone; semaglutide; Pentoxifylline; baricitinib

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, open-label, parallel-group, clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Active Comparator): Maximally tolerated dose of ACEi or ARB (but not both), SGLT2i, and finerenone. Blood pressure target <130/80 mm Hg
  Interventions: Drug: ACEi / ARB, SGLT2i, finerenone, semaglutide, pentoxifylline, hydrochlorthiazide, baricitinib
- Albuminuria-reduction protocol (Experimental): Maximally tolerated dose of ACEi or ARB (but not both), SGLT2i, and finerenone. Thereafter addition of semaglutide, pentoxifylline, hydrochlorothiazide, and baricitinib.
  Blood pressure target <130/80 mm Hg, but if still UACR >300 further reduction in blood pressure will be attempted as tolerated.
  Interventions: Drug: ACEi / ARB, SGLT2i, finerenone, semaglutide, pentoxifylline, hydrochlorthiazide, baricitinib

INTERVENTIONS:
Drug: ACEi / ARB, SGLT2i, finerenone, semaglutide, pentoxifylline, hydrochlorthiazide, baricitinib — Standard of care for diabetic kidney disease.

SUMMARY:
The purpose of this trial is to investigate the feasibility and safety of implementing a protocol-based treatment aggressively targeting albuminuria in subjects with biopsy-proven diabetic nephropathy and severely elevated albuminuria. If this approach is feasible, the results of the trial will inform the design of a large-scale randomized clinical trial to evaluate the effect of this treatment on hard kidney endpoints (initiation of dialysis, kidney transplantation, and death from kidney failure) in subjects with biopsy-proven diabetic nephropathy and severely elevated albuminuria.

DETAILED DESCRIPTION:
Diabetic kidney disease (DKD) is the leading cause of end-stage kidney disease (ESKD) worldwide and declining kidney function is associated with a graded increase in the risk of death or hospitalization. Thus, prevention of kidney disease progression is of vital importance to prevent excess morbidity and mortality among people with DKD.

Increasing levels of albuminuria in patients with DKD are associated with a graded increase in the risk of developing ESKD and among patients with nephrotic-range albuminuria (i.e. > 2.000 mg/day) progressive decline in kidney function is particularly rapid. The currently available drugs which have demonstrated delayed progression to ESKD in DKD (captopril, losartan and irbesartan, canagliflozin, dapagliflozin, empagliflozin, and finerenone) all reduce albuminuria independently of blood pressure reductions, but it has long been debated whether reductions in albuminuria by itself reflects a reduction in the risk of ESKD or whether this is simply a by-product of treatment. Whether interventions targeting reductions in albuminuria reduce the incidence of ESKD has not been formally tested in a randomized controlled trial of hard kidney endpoints (e.g. initiation of dialysis, kidney transplantation or death from kidney disease).

We wish to conduct a randomized controlled trial in which we will test whether an aggressive treatment strategy of lowering albuminuria reduces the incidence of hard kidney endpoints compared to standard-of-care among patients with nephrotic-range albuminuria and very high risk of progression to ESKD. However, prior to conducting such a trial it is necessary first to test whether it is even possible to sufficiently lower albuminuria by these means. Therefore, we wish to first conduct a pilot trial to investigate the feasibility of such an approach.

Participants will be randomized 1:1 to standard-of-care or an albuminuria-reduction protocol. In the albuminuria-reduction protocol, subjects will be treated with various drugs that have all been shown to reduce albuminuria in DKD (although not all have been shown to reduce hard kidney outcomes). At each monthly study visit, drugs will be added or withdrawn in an attempt to maximally reduce albuminuria. Drugs that reduce albuminuria by <10% since the last study visit will be discontinued. Drugs that successfully reduce albuminuria by >10% will be continued and further drugs will be added.

After 9 months subjects will discontinue protocol drugs and resume their previous medical care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of diabetes mellitus type 2 (American Diabetes Association / European Association for the Study of Diabetes (ADA/EASD) definition)10
* Biopsy-proven diabetic nephropathy
* UACR ≥ 2,000 mg/g or
* UACR ≥ 1,500 mg/g if treated with sodium-glucose cotransporter 2 inhibitor (SGLT2i)
* Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73 m2
* Negative pregnancy test and use of highly effective and safe contraception
* Able to give informed consent.

Exclusion Criteria:

* Kidney transplant recipient
* Findings on kidney biopsy suggestive of other or concomitant glomerulonephritis (findings associated with hypertensive nephropathy are not exclusion criteria).
* Plasma potassium at baseline > 5.2 mmol/L.
* Active malignancy (basal or squamous cell skin carcinoma, localised prostate cancer, and cancer with no signs of reoccurrence after 5 years are exempt from this).
* Systolic heart failure with NYHA class III-IV.
* Liver failure classified as Child-Pugh C.
* Primary hyperaldosteronism.
* Previous cerebral or retinal haemorrhage.
* Biliary obstructive disorders.
* Acute myocardial infarction within the last three months.
* Severe cardiac arrhythmias.
* Clinically active gout.
* Plasma sodium at baseline < 135 mmol/L.
* Other diseases or conditions, which, in the opinion of the site investigator, would prevent participation in or completion of the trial.
* Treatment with potent CYP3A4 inhibitors.
* Participation in other interventional trials.
* Allergy towards one of more of the drugs to be used during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
urine albumin/creatinin-ratio (UACR) reduction to less than 50% of baseline | after 9 months of treatment
  number of subjects achieving this endpoint

SECONDARY OUTCOMES:
UACR reduction to less than 70% of baseline | after 9 months of treatment
  number of subjects achieving this endpoint
UACR less than 300 | after 9 months of treatment
  number of subjects achieving this endpoint
difference in UACR | after 9 months of treatment
  between-groups difference in UACR
difference in UACR | after 10 months of treatment (1 month off study drugs)
  between-groups difference in UACR
difference in eGFR | after 9 months of treatment
  between-groups difference in eGFR
difference in eGFR | after 10 months of treatment (1 month off study drugs)
  between-groups difference in eGFR
difference in systolic and diastolic blood pressure | after 9 months of treatment
  between-groups difference in blood pressure
difference in systolic and diastolic blood pressure | after 10 months of treatment (1 month off study drugs)
  between-groups difference in blood pressure
incidence of plasma potassium >5.5 mmol/L | after 9 months of treatment
  number of subjects achieving this endpoint
incidence of plasma potassium >6.0 mmol/L | after 9 months of treatment
  number of subjects achieving this endpoint
incidence of symptomatic hypotension | after 9 months of treatment
  number of subjects achieving this endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Iain Bressendorff, MD PhD, Principal Investigator — Herlev and Gentofte Hospital
Locations (1):
- Department of Nephrology, Herlev and Gentofte Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No